CLINICAL TRIAL: NCT01945125
Title: Effects of Thyroid Hormone Withdrawal and Recombinant Human Thyroid Stimulating Hormone in Glomerular Filtration Rate During Radioiodine Therapy
Brief Title: Effects of THW and rhTSH in Glomerular Filtration Rate During RIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NP97/10
Record Dates: First submitted 2013-09-09; First posted 2013-09-18 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2013-11

CONDITIONS: Other Impaired Renal Function Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- THW Group (No Intervention): Patients under THW stimulation for RIT
- rhTSH Group (Other): Patients under rhTSH stimulation for RIT
  Interventions: Other: rhTSH Group

INTERVENTIONS:
Other: rhTSH Group — Patients receiving rhTSH for RIT stimulation
  Arms: rhTSH Group

SUMMARY:
To observe the influence of thyroid hormone withdrawal and of recombinant human TSH during radioiodine therapy in renal function.

DETAILED DESCRIPTION:
Radioiodine therapy in thyroid carcinoma is a procedure performed for over six decades, and there is a vast literature in respect of its value in the complementary treatment of this neoplasia. This procedure also promotes a reliable follow-up based on sequential thyroglobulin dosages and makes possible to reduce the disease recurrence rate. One of the main aspects of the patients preparation before receiving the radioiodine consists in promoting stimulation for an effective uptake of the radioiodine, obtained either by endogenously TSH level elevation after post-surgical thyroid hormone withdrawal, or exogenously after use of recombinant human TSH. This last alternative does not demand suspension of thyroid hormone reposition after total thyroidectomy. Although not fully comprehended, it is known that hypothyroidism results in renal function hazard, which is reverted after hormonal reposition. It is also known that renal function modifies the radioiodine residence time and that the longer this time, the greater the patient's radiation exposure will be, and consequently with undesired irradiation of healthy tissues and organs. So theoretically stimulating the patient with recombinant human TSH could avoid the transient deficient renal function, promoting a lower radioiodine residence time and consequently lowering radiation exposure in this therapy.

This project aims to evaluate the effects of the different stimulation, endogenous and exogenous, over renal function by glomerular filtration rate determined by 51Cr-EDTA. This will be a controlled and randomized study in which 44 patients that has clinical indication of remnant ablative radioiodine treatment will be prepared by either one of the TSH stimulation procedures. Additionally radiation dosimetry calculus will be done to analyze the levels of the patient's radiation exposure associated with each of the uptake stimulation procedures for radioiodine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Normal Renal Function

Exclusion Criteria:

* Abnormal Renal Function
* Renal metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Observation of differences in glomerular filtration rate with THW or rhTSH in radioiodine therapy | participants will be followed during radioiodine treatment, from the decision of treatment to the post treatment whole body scan, an expected average of 2 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: George B Coura Filho, MD, Principal Investigator — ICESP-FMUSP
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Coura-Filho GB, Willegaignon J, Buchpiguel CA, Sapienza MT. Effects of Thyroid Hormone Withdrawal and Recombinant Human Thyrotropin on Glomerular Filtration Rate During Radioiodine Therapy for Well-Differentiated Thyroid Cancer. Thyroid. 2015 Dec;25(12):1291-6. doi: 10.1089/thy.2015.0173. Epub 2015 Nov 5. PMID 26446582